CLINICAL TRIAL: NCT06370455
Title: Comparison of Septal Advancement Flap and Columellar Strut in Preserving, Restructuring, and Reshaping the Nasal Tip Contour in Rhinoplasty
Brief Title: Comparison of Septal Advancement Flap and Columellar Strut Effect on Nasal Tip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaied Allam, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 36264MS429/11/23
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Rhinoplasty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Septal advancement flap group (Active Comparator): Fifteen patients will undergo septal advancement flap technique The mucoperichondrial flaps are elevated over the cartilaginous septum and the caudal perpendicular plate of the ethmoid. investigator will take L shape flap of the dorsal and anterior end of cartilaginous septum then advance them and suture the flap at certain points so can support the nasal tip.
  Interventions: Procedure: comparison of septal advancement flap effect on nasal tip in primary rhinoplasty to columellar strut technique
- Columellar strut group (Active Comparator): fifteen patients will undergo columellar strut technique. investigator will extract columellar strut from septal cartilage then insert it between the two medial crura n the intercrural space and sutured to nasal spine so can support nasal tip.
  Interventions: Procedure: comparison of septal advancement flap effect on nasal tip in primary rhinoplasty to columellar strut technique

INTERVENTIONS:
Procedure: comparison of septal advancement flap effect on nasal tip in primary rhinoplasty to columellar strut technique — All patients will be operated on under general anesthesia through an open rhinoplasty then will undergo 2 different procedures according to each group.

SUMMARY:
The aim of the study to compare and evaluate the effect of septal advancement flap in preserving and reshaping the nasal tip with columellar strut graft

DETAILED DESCRIPTION:
The ideal tip support graft should support the exact position over time, avoid stiffness of a natural soft structure of the tip, be easily harvested typically septal cartilage, facilitate surgeon control of rotation and projection.

To address these desirable features the septal advancement flap (SAF) was developed. The septal advancement flap (SAF) is a rotational advancement flap of the superior and caudal aspects of the cartilaginous septum that enables the surgeon to create stable and accurate tip shape and position. This is a technically easy and reliable flap mainly applicable to primary rhinoplasty.

so investigator compare between this new technique and old one like columellar strut to know the effect on nasal tip

ELIGIBILITY:
Inclusion Criteria:

* Droopy nasal tip

Exclusion Criteria:

* severely deficient cartilaginous septum.
* previous nasal operations, history of cleft lip or cleft palate.
* bleeding disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-08-23 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
subjective assessment using Rhinoplasty Outcome Evaluation Questionnaire | preoperative and one month postoperative
  Assessment of patient satisfaction with primary septorhinoplasty using the Arabic Rhinoplasty Outcome Evaluation (ROE) Questionnaire and comparing the preoperative with postoperative scores. The ROE comprises 6 questions. Each answer is scored on a scale from 0-4, where 0 corresponds to the "most negative answer" and 4 corresponds to the "most positive answer." As a result, the total score can range from 0 to 24.
  To make the results easier to understand, the total score can be divided by 24 and multiplied by 100 to obtain a value between 0% and 100%, where higher values represent greater patient satisfaction.
measuring the degree of tip projection and rotation preoperative and postoperative | Preoperative,one month and six months postoperative
  Objective assessment by measuring the degree of tip projection and rotation preoperative and postoperative by using the angle between the columella and the line intersecting the junction between the columella and the upper lip and the vermilion border of the upper lip for measuring the nasolabial angle.

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngology department -Tanta University Hospitals, Tanta, Egypt

REFERENCES:
- [Background] Goncalves Ferreira M. Septal Advancement Flap: Preserving, Restructuring, and Reshaping the Nasal Tip Contour with a Novel Flap. Facial Plast Surg Aesthet Med. 2023 Jul-Aug;25(4):279-284. doi: 10.1089/fpsam.2023.0060. Epub 2023 Apr 10. PMID 37036815